CLINICAL TRIAL: NCT01601730
Title: Combination Therapy With Modafinil and Escitalopram for the Treatment of Cocaine Dependence
Brief Title: Modafinil - Escitalopram Study for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-25669; 1RC1DA028387 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-12-10; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Cocaine Dependence; Cocaine Abuse; Cocaine Addiction; Substance Abuse
Keywords: Cocaine; Modafinil; Escitalopram
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Modafinil; Escitalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Modafinil 200 mg + Escitalopram 20 mg (Active Comparator)
  Interventions: Drug: Modafinil and Escitalopram
- Modafinil 200 mg (Active Comparator)
  Interventions: Drug: Modafinil
- Escitalopram 20 mg (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Modafinil and Escitalopram — Treatment 4: Modafinil 200 mg + Escitalopram 20 mg
  Other Names: Provigil; Lexapro
  Arms: Modafinil 200 mg + Escitalopram 20 mg
Drug: Placebo — Matching oral placebo capsules as control (Treatment 1: Modafinil 0 + Escitalopram 0).
  Other Names: Sugar pill
  Arms: Placebo
Drug: Modafinil — Treatment 2: Modafinil 200 mg + Escitalopram 0.
  Other Names: Provigil
  Arms: Modafinil 200 mg
Drug: Escitalopram — Treatment 3: Modafinil 0 + Escitalopram 20 mg.
  Other Names: Lexapro
  Arms: Escitalopram 20 mg

SUMMARY:
The purpose of this study is to improve the efficacy of modafinil as a potential treatment for cocaine dependence.

DETAILED DESCRIPTION:
In this application, we propose an augmentation strategy intended to improve the efficacy of modafinil as a potential treatment for cocaine dependence. Recent data indicates that during chronic treatment modafinil produces substantial dopamine transporter (DAT) inhibition. Given that cocaine inhibits DA, norepenepherine (NE) and serotonin (5-HT) reuptake, it is highly likely that targeting more than one neurotransmitter system will be necessary for a medication to be effective. Assuming that this statement is true, we hypothesize that a combination pharmacotherapeutic approach that concurrently modulates multiple neurotransmitter systems will likely demonstrate a clinically significant level of efficacy above trials in which a single medication is used. The proposed approach is based on preclinical data indicating that medications that increase brain 5-HT levels reduce the effects of stimulants. We hypothesize that combining modafinil with a selective serotonin reuptake inhibitor (SSRI), which will increase synaptic levels of 5-HT, will further improve the efficacy of modafinil for reducing the effects produced by cocaine.

Specific Aims: 1) to determine the effects of treatment with oral modafinil (0 or 200 mg) plus the SSRI escitalopram (0 or 20 mg) on the subjective and reinforcing effects produced by intravenous cocaine (0 and 20 mg) in the laboratory. 2) to characterize the cocaine dependent population and the genetic basis for the rewarding effects produced by cocaine. 3) to characterize the effect of both modafinil treatment and cocaine exposure onBrain Derived Neurotrophic Factor (BDNF) in plasma. We hypothesize that both modafinil treatment and cocaine exposure will alter plasma levels of BDNF. 4 a) provide a more frequent measure of heart rate (15 sec vs. 5 minutes) and b) measure a new dependent variable, physical activity, on days with and without cocaine exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Be a cocaine-dependent volunteer who is non-treatment-seeking.
2. Meet DSM-IV criteria for cocaine dependence as determined by SCID or MINI, and has provided at least one cocaine-positive urine specimen within the 2 weeks prior to enrollment.
3. Be male or female, between 18 - 55 years old.
4. Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
5. Female subjects must be non-nursing and postmenopausal, have had a hysterectomy, undergone tubal ligation, or have a negative pregnancy test and agree to use birth control.
6. Has medical history, physical exam, and screening laboratory results that demonstrate no contraindication to participation.
7. Be experienced with smoking or i.v. use as a route of cocaine administration.

Exclusion Criteria:

1. Has a history of a medical adverse reaction to cocaine or other psychostimulants, including loss of consciousness, chest pain, cardiac ischemia, or seizure.
2. Has a current psychiatric disorder other than cocaine abuse or dependence (e.g., major depression, bipolar disorder, schizoaffective disorder, schizophrenia).
3. Meets DSM-IV criteria for dependence on other illicit drugs (e.g., methamphetamine, heroin).
4. Has received opiate-substitution therapy within 2 months of enrollment.
5. Has a current or past history of seizure disorder, including alcohol- or psychostimulant- related seizures, febrile seizures, or family history of seizure disorder.
6. Has a diagnosis of adult asthma, or chronic obstructive pulmonary disease, including a history of acute asthma within the past two years, and those with current or recent (with the past two years) treatment with an inhaled or oral b-adrenergic agonist.
7. Has had head trauma that resulted in neurological sequelae (e.g., loss of memory for greater than 5 min or that required hospitalization).
8. Has an unstable medical condition, which, in the judgment of investigators, would make participation hazardous, including, but not limited to, AIDS, acute hepatitis, active TB, unstable cardiac disease, unstable diabetes, hepatic or renal insufficiency (serum bilirubin or creatinine exceeding 1.5 the upper limit of normal, respectively).
9. Be pregnant or lactating (nursing), or a fertile woman not practicing adequate methods of contraception or planning to become pregnant within one month of conclusion of the study.
10. Has a history of suicide attempts within the past year and/or current suicidal ideation/plan.
11. Has clinically significant ECG abnormalities, including QTc interval prolongation >450 ms in men or >480 ms in women.
12. In the opinion of the PI, be expected to fail to complete the study protocol due to probable incarceration or relocation from the clinic area.
13. Has clinically significant laboratory values (outside of normal limits), in the judgment of the PI.
14. Is currently taking SSRIs, monoamine oxidase inhibitors or pimozide.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The effects of modafinil and/or escitalopram and cocaine on cardiovascular measures
  Before and after each cocaine infusion, physiologic responses will be closely monitored using repeated HR, BP, and ECG readings. To evaluate safety, a DSMB will meet annually and following any serious AE to examine data as well as any new published information on modafinil and/or escitalopram relevant to the project. The number of AEs (including arrhythmias and ECG changes), changes in BP and HR, changes in cocaine PKs, and changes in mood and psychiatric symptoms (using the BSI, BDI, POMS, and BPRS) will also be assessed throughout the study.

SECONDARY OUTCOMES:
The effects of modafinil and/or escitalopram and cocaine on subjective measures
  The ability of modafinil and/or escitalopram, as compared to placebo, to reduce cocaine-induced craving will be measured by VAS and ARCI.
The effects of modafinil and/or escitalopram on reinforcing effects produced by cocaine
  The ability of modafinil and/or escitalopram, as compared to placebo, to reduce reinforcing effects produced by cocaine will be measured by choices for cocaine vs. money in the self-administration assay.

CONTACTS AND LOCATIONS:
Overall Officials: Richard De La Garza, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States